CLINICAL TRIAL: NCT07185919
Title: Registry to Document Treatment Effectiveness, Safety, Including Prospective Long-term Outcomes in Participants With Progressive Familial Intrahepatic Cholestasis (PFIC) Who Take Odevixibat (Bylvay)
Brief Title: A Study of the Effectiveness, Safety and the Long-term Outcomes of Participants With Progressive Familial Intrahepatic Cholestasis (PFIC) Who Take Odevixibat (Bylvay) in South Korea
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60240-030
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will collect information from people with Progressive Familial Intrahepatic Cholestasis (PFIC) as they use odevixibat in their daily lives. Odevixibat is a medicine that helps people with PFIC, a type of rare disease that makes their liver not work well and causes itching and yellow skin. Odevixibat was first allowed to be used for PFIC in babies older than 6 months by the European Medicines Agency (EMA) on 16 July 2021 and by the United States Food and Drug Administration (FDA) on 20 July 2021 for itching in babies older than 3 months. Obevixibat was approved by the Ministry of Food and Drug Safety (MFDS) in South Korea on 23 August 2024.

This study will collect information to see how well and how safe odevixibat is in the long run for participants in South Korea.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with PFIC (all types) who have been prescribed odevixibat (independently of the decision to enrol the participant in this registry) by their treating physician
2. On (or starting) active odevixibat treatment Note: Participants can remain in the registry during odevixibat treatment interruptions

Exclusion criteria:

1. Currently participating in a clinical trial with odevixibat
2. Currently participating in any interventional clinical trial for PFIC
3. Have any contraindication to odevixibat as per the approved label in South Korea.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry population will comprise participants with PFIC (all types) enrolled into the Ipsen odevixibat PFIC registry. Participants with PFIC who have been prescribed odevixibat by their treating physician will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing Adverse Events (AEs) | From first ICF signature and up to end of data collection (approximately 7 years of data collection)
  An Adverse event (AE) is any untoward medical occurrence, temporally associated with the use of study intervention, whether or not related to the study intervention.

SECONDARY OUTCOMES:
Event-free survival (EFS) | From first ICF signature and up to end of data collection (approximately 7 years of data collection)
  EFS is defined as time from the start of odevixibat treatment to the first occurrence of surgical biliary diversion, liver transplant, or death
Surgical biliary diversion-free survival | From first ICF signature and up to end of data collection (approximately 7 years of data collection)
  Surgical biliary diversion-free survival is defined as time from the start of odevixibat treatment to the first occurrence of surgical biliary diversion or death
Liver transplant-free survival | From first ICF signature and up to end of data collection (approximately 7 years of data collection)
  Liver transplant-free survival is defined as time from the start of odevixibat treatment to the first occurrence of liver transplant or death
Overall survival (OS) | From first ICF signature and up to end of data collection (approximately 7 years of data collection)
  OS is defined as the time from the start of odevixibat treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/